CLINICAL TRIAL: NCT04914624
Title: Effects of Different Physical Therapy Programs on Pulmonary Rehabilitation in Patients With Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hao Long, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-ZJD-001
Record Dates: First submitted 2020-12-30; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Rehabilitation
Keywords: pulmonary rehabilitation; external diaphragm pacemaker; expiratory pressure therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular ACBT training (Placebo Comparator): Including quitting smoking, ACBT training, cough practicing.
  Interventions: Behavioral: ACBT training
- Positive expiratory pressure therapy (Experimental): Use acpella®PEP therapeutic system and regular nursing care.
  Interventions: Device: acpella®PEP
- External diaphragm pacemaker (Experimental): Patients are trained to use external diaphragm pacemaker and receive regular nursing care.
  Interventions: Device: EDP-type II external diaphragm pacemaker

INTERVENTIONS:
Behavioral: ACBT training — Performed 5 days before surgery and one month after surgery, twice a day.
  Arms: Regular ACBT training
Device: acpella®PEP — Continuously instruct patients to perform positive expiratory pressure training 5 days before surgery and one month after surgery, twice a day.
  Arms: Positive expiratory pressure therapy
Device: EDP-type II external diaphragm pacemaker — Use external diaphragm pacemaker to stimulate patients' diaphragms.
  Arms: External diaphragm pacemaker

SUMMARY:
This study applies external diaphragm pacemaker and positive expiratory pressure therapy to patients who received thoracic surgeries, in order to explore the effects of different physical therapy programs on pulmonary rehabilitation in patients with lung cancer. As well as we hope that these physical training programs can effectively improve the lung function of patients, reduce postoperative pulmonary complications, hospitalization days, hospitalization expenses, etc.

DETAILED DESCRIPTION:
This study applies external diaphragm pacemaker and positive expiratory pressure therapy to patients who received thoracic surgeries, ninety patients may be enrolled in this study.

Some metrics are used to evaluate the pulmonary rehabilitation status in postoperative patients which include pulmonary function test, 6-Min Walking Test，Borg index, complications incidence, chest tube draining time, and diaphragm muscle mobility.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with non-small cell lung cancer with clear pathological cytology by fiberoptic bronchoscopy and CT, and plan to undergo lobectomy or segmentectomy under general anesthesia for tracheal intubation;
2. Age 18-80 years old;
3. Those who have stable vital signs and can participate in this research;
4. Pulmonary function test FEV1/FVC>0.8.
5. Volunteer to participate in this research and sign an informed consent form.

Exclusion Criteria:

1. Pneumonectomy patients;
2. Wedge resection patients
3. Patients with distant metastasis of cancer;
4. Patients with other malignant tumors;
5. Severe complications occurred during the operation, and respiratory function training and testing are not allowed before and after Evaluator;
6. Patients with severe physical or mental illness who cannot cooperate with the test;
7. Patients with pacemakers, active tuberculosis, and pneumothorax.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline Forced Expiratory Volume In One Second at one month after surgery | baseline (before the surgery), and one month after surgery
  Evaluate the change of Forced Expiratory Volume In One Second before the surgery and one month after surgery by conducting Pulmonary Function Test on resectable NSCLC patients

OTHER OUTCOMES:
The change from baseline Borg Score at one month after surgery. | baseline (before the surgery), and one month after surgery
  Borg Score is a rating of perceived exertion which is a reliable indicator to monitor and guide exercise intensity.It allows individuals to subjectively rate their level of exertion during exercise testing.We would record patients' Borg Score after 6 minutes walking test
Complications incidence | One month after surgery
  Record the complications of patients after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat sen University cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen X, Li C, Zeng L, Rong T, Lin P, Wang Q, Guo Z, Long H, Zhong J. Comparative efficacy of different combinations of acapella, active cycle of breathing technique, and external diaphragmatic pacing in perioperative patients with lung cancer: a randomised controlled trial. BMC Cancer. 2023 Mar 28;23(1):282. doi: 10.1186/s12885-023-10750-4. PMID 36978035